CLINICAL TRIAL: NCT07343700
Title: Community Expecting: Exercise During Pregnancy for Sedentary Women With Obesity
Brief Title: Community Expecting: Exercise During Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Taren Swindle, Associate Professor, Arkansas Children's Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 297995
Record Dates: First submitted 2025-12-04; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Physical Activities
Keywords: Pregnancy; Prenatal Exercise; Prenatal fitness; Community; Implementation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): In the intervention group, women exercise in small groups with a certified personal trainer who has passed a certification process related to the research and exercise protocol. Specifically, women in the intervention are asked to work out three times per week, progressing to 45 minutes each session within the first 6 weeks. Participant workouts are focused primarily on body weight exercises although participants also receive resistance bands for use in the workouts. Participants can choose to watch a recorded workout rather than attend a live session for 1 of their 3 workouts for the week.
  Interventions: Behavioral: Community Expecting
- Control (No Intervention): Women receive standard care and encouraged to follow doctor's recommendations for physical activity

INTERVENTIONS:
Behavioral: Community Expecting — our team adapted EXPECTING for community delivery through extensive input from prior participants and community advisors using an implementation science framework. In our prior project plan, the EXPECTING intervention was successfully adapted to community settings and tested for its acceptability, feasibility and fidelity using the Replicating Effective Programs (REP) strategy8 with input from diverse community partners. This process resulted in 4 key adaptations to define the COMMUNITY EXPECTING Intervention and 3 implementation strategies to support its uptake in the community. Dose, frequency, type, and targeted exertion during exercise were retained as core components from the original EXPECTING study. All intervention components have been tested in the community.
  Arms: Exercise

SUMMARY:
Regular physical activity during pregnancy is safe and offers many health benefits for both mothers and their babies. Research over the past decade shows that exercise can help pregnant women gain a healthy amount of weight, lower their risk of gestational diabetes and high blood pressure, and reduce stress, anxiety, and symptoms of postpartum depression. Babies also benefit when their mothers are active, with lower risks of preterm birth, unhealthy birth size, and childhood obesity.

Despite this strong evidence, very few exercise programs for pregnant women have been tested in real-world community settings, such as fitness centers, community health programs, or local organizations. Even fewer studies explain how these programs were delivered or what helped them succeed. Without this information, it is difficult for communities and health programs to offer exercise support that is both effective and practical for pregnant women.

To address this gap, the research team adapted an evidence-based program called EXPECTING so it could be delivered by community organizations. Previous participants and community advisors helped to understand what changes were needed to make the program easier to offer while still keeping it safe and effective. The core parts of the program, including the type, amount, and intensity of aerobic and strength-building exercises, remained the same and are based on established pregnancy exercise guidelines.

The adapted program, called COMMUNITY EXPECTING, includes both aerobic exercise and resistance training. The research team also developed specific supports to help community instructors deliver the program consistently and with confidence. All program components have already been tested in community settings and shown to be realistic, acceptable, and delivered as planned.

This study will examine whether offering a structured exercise program in community settings helps pregnant women be more physically active than usual prenatal care alone. We will also assess whether the program can be delivered successfully and in a way that works for both participants and community providers. The results will help determine whether COMMUNITY EXPECTING is a practical approach for supporting healthy pregnancies in real-world settings.

DETAILED DESCRIPTION:
In the COMMUNITY EXPECTING intervention, women exercise in small groups with a certified personal trainer who has passed a certification process related to the research and exercise protocol. Specifically, women in the COMMUNITY EXPECTING intervention are asked to work out three times per week, progressing to 45 minutes each session within the first 6 weeks. Participant workouts are focused primarily on body weight exercises although participants also receive resistance bands for use in the workouts. Participants can choose to watch a recorded workout rather than attend a live session for 1 of their 3 workouts for the week. Participants will be provided with postpartum support, and incentive schedule that will promote scalability and sustainability.

Additional details of the program include the following:

1. Participants will be asked to complete at least 2 live, in-person (i.e., synchronous) training sessions per week; the third session can be via a Docebo workout. Docebo may also be used in inclement weather. Participants in the exercise group can access recorded workouts on the Docebo learning platform for participants (https://www.communityexpecting.com/learn). Docebo is a secure and HIPPA compliant platform where participants can use multiple video platforms (e.g., zoom, Teams) to have live training sessions with a trainer and access recorded training sessions. Participants in the exercise group will receive training in the use of Docebo and have support from the research team to navigate all components. We may also house content on UAMS web pages as needed.
2. Participants can elect to have one person join them for the workout sessions. Each person participating in the workouts that is not a study participant will sign and return the "Workout "Buddy" Release and Waiver of Liability Form," approved by ACH legal representatives.
3. All trainers will receive a 3-hour training in the protocol and receive 80% or higher on a knowledge assessment post-training before being certified to provide training for the study. We will train the certified personal trainers to deliver the sessions with fidelity to the intended format using body weight exercise and minimal equipment (e.g., resistance band). Trainers will be required to submit videos of sessions or agree to live observations for fidelity scoring to the research team.
4. The workouts will include 3 major components: (1) Aerobics, (2) Resistance Training, and (3) Stretching. Aerobic activities will be done primarily without equipment; examples include walking, marching in place, low impact jumping jacks (side step with overhead jack). If participants have access to equipment (e.g., treadmill, swimming pool), only low-impact activities will be included. Resistance activities are designed to strengthen major muscle groups except for the abdominals. Target muscle groups include arms, chest, back, hips/glutes, and legs. These activities will use bodyweight and/or resistance bands (e.g., upper body rows, seated leg curls). Stretching activities are aimed to increase flexibility and mobility of the whole body (e.g., calf stretches, gentle neck stretches). Table 1 details the duration of each activity across the weeks of the intervention. Workouts will occur 3 times per week until delivery or a contraindication for exercise (e.g., doctor's request). The goal is for the aerobic and resistance training to be of moderate intensity. The trainer will monitor the intensity of the workout by asking the participant to rate their perceived exertion during the workouts and using the "talk test" to ensure the participants can speak short sentences without difficulty. Perceived exertion is rated using an established measure - the Rate of Perceived Exertion (RPE) scale, which is rated on a scale of 6 -20. The target for participants for aerobic and resistance components is 12-14. The trainers will suggest modifications to ensure moderate intensity (e.g., slowing/increasing pace, adding/decreasing resistance). There is no intensity target for the stretching portion of the sessions. Following each workout, participants will complete a short survey acknowledging their attendance at the workout, average heart rate during the workout, and their RPE following the session. Surveys are completed and data stored using REDCap.
5. After delivery and clearance for exercise from their doctor, mothers will have the option to continue with the program for up to 12 months. If participants elect to receive post-partum support, they could be in the study up to 18 months. This post-partum program will support mothers' re-entry into exercise when/if desired.

   * "The study was registered once the requirement for registration in an ICMJE-accepted registry was identified. No changes were made to study procedures or participant activities as a result of this timing

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Having a BMI ≥ 30
* Not currently meeting guidelines for 150 min of moderate physical activity per week.
* All children born to mother participants will be included and eligible.

Exclusion Criteria:

* Non-English speaking individuals.
* Contraindications for exercise (preeclampsia-eclampsia, premature rupture of the membranes, antepartum hemorrhage, placenta previa, or multiple gestation),) as determined by the investigators to affect the outcomes of interest
* Using recreational drugs, tobacco, or alcohol during their pregnancy.
* < 11 or > 16 weeks gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Step Logs | Weekly from enrollment (baseline) through delivery, assessed throughout pregnancy (up to ~40 weeks gestation).
  All "expecting mother" participants in both groups will receive a FitBit arm bracelet to self-monitor activity levels and for the research team to monitor their physical activity levels. They will also submit their step counts on a weekly basis and/or give permission for us to access their step count data from the Fitbit records. Weekly step count logs are sent to the participant through REDCap via email or text message. The message contains a "survey link" produced by REDCap, where the participant reports step count data or answers survey questions. Upon completion, the data is automatically upload to REDCap for later analysis.

SECONDARY OUTCOMES:
Maternal Health Assessment | Assessed at baseline (post-consent), during the third trimester of pregnancy, 6 -12 weeks postpartum, and 1 year postpartum (as close as possible but can exceed).
  To obtain both mother anthropometrics and vital signs, we will use the Health Assessment forms via healthcare providers and provide our community workout locations with equipment to collect height, weight, and blood pressure of mothers if there are barriers to collecting this information from the healthcare provider. Health assessments will be collected from expecting mother participants in both groups.
Beck Depression Inventory | At enrollment (pre-third trimester), during the third trimester, at 6 weeks postpartum, and at 1 year postpartum.
  Expecting mother participants in both groups will complete this measure. Maternal signs and symptoms of depression will be evaluated using the Beck Depression Inventory-II (BDI-II) The BDI-II is a 21-item self-report questionnaire, rated on a four-point scale, which has been validated for use in pregnancy (37). Each item consists of four statements, scored 0-3, and total scores can range from 0 to 63. The BDI-II will be analyzed to determine if there is any evidence of changes in depression signs and symptoms during pregnancy and postpartum and determine if any relationship exists with changes in physical activity. The BDI-II will be sent to the participant via a survey link through REDCap via email or text and they will fill out the questionnaire, which will be saved in REDCap. This information is being collected because mental health may be an important moderator of the intervention's effects.
Trainer fidelity | Weekly at site or cohort launch, followed by monthly fidelity assessments during the intervention period (up to ~12 months).
  Study team members will monitor fidelity to implementation of delivery. This will be completed in-person or via video recorded submissions from community sites. The fidelity assessment by a study team member of the community-based trainer will be completed in person or virtually. Feedback will be shared in a timely fashion with trainers as needed to correct any deviations from the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Taren Swindle, Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Research Institute, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No